CLINICAL TRIAL: NCT02043249
Title: Cord Milking and Activity Of The Immune System In Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HYMC 0042-13
Record Dates: First submitted 2013-11-13; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2013-11

CONDITIONS: Preterm Delivery
Keywords: DELAYED CORD CLAMPING; MILKING OF CORD; PREMATURE INFANTS; LEVEL OF IgG IN NEONATES
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CORD MILKING (No Intervention): WITHOUT MILKING
  Interventions: Other: CORD MILKING

INTERVENTIONS:
Other: CORD MILKING — MILKING OF UMBILICAL CORD OF THE BABY
  Other Names: UMBLICAL MILKING

SUMMARY:
In the embry life there is a passage of IgG type, from the mother to tha embryoyo and only in the age of 3-5 month after birth the infant start to develop them by himself.

In preterm infants the starting point of the level of the IgG's is lower from the level of term infants.

Delayed cord clamping /milking it was prooved in many researches as benificial in terms of : levels of hemoglobin; hematocrit and feritin in the neonats. Also benefits were proved by means of less need for blood tranfusion, less intra ventricular hemorrhage; necrotzing entero colitis and iron deficiency anemia. The hypothesis is that delayed clamping /milking it will increse the level of IgG's in preterm infants. The end point hypothesis is that delayed cord clamping /milking cause to less fever disease or hospitalization it the neonats.

DETAILED DESCRIPTION:
In this study we come to a prove that if we miking the cord in preterm infats we will increse the level of IgG .

ELIGIBILITY:
Inclusion Criteria:

* PRETERM INFANS BETWEEN 24+0/7 TO 36

  * 6/7 WEEKS.
  * NEWBORN FOR MOTHER WHO AGREE TO PARTICIPATE IN THE RESEARCH WHO DELIVER IN NORMAL DELIVERY / PLANED OR URGENT CESARIAN DELIVERY

Exclusion Criteria:

* INTRA UTERINE GROWTH RESTRICTION, INFANT UNDER 10% TO AGE OF PREGNANCY.
* MOTHER WHO IS NOT WILLING TO PARTICIPATE IN RESEARCH.
* NEONATES TO MOTHER WHOM SUSPECTED TO BE IMMUNO- COMPROMISED OR HAVING INFECTION AROUND DELIVERY.

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
levels of IgG in preterm infats | 24 hours after delivery and after 24 hours..
  Blood test for IgG's level from the baby in :
  at delivery . 24 hours after delivery. before discharg from hospital

SECONDARY OUTCOMES:
Mother's telephone questioning about the infant disease: fiver / hospitalization/tretment wit antibiotic. | 3 and 6 month after delivery
  Phone call interview of the mother in 3 and 6 month from delivery about : emergengy room admission; hospitalization, fever disease and antibiotic treatment in this time period.

CONTACTS AND LOCATIONS:
Overall Officials: Rivka Frenkel, MD, Principal Investigator — Hellel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel